CLINICAL TRIAL: NCT02351388
Title: Ameliorating Depression in Alzheimer's Disease Patients by Transcranial Direct Current Stimulation (ADAPT) - Preliminary Research
Brief Title: Transcranial Direct Current Stimulation for Depression in Alzheimer's Disease Patient - Preliminary Research
Acronym: ADAPT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: failure to recruit enough number of participants
Sponsor: National Center of Neurology and Psychiatry, Japan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A2014-086
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Alzheimer Disease; Depression
Keywords: Alzheimer's disease; Depressive symptoms; Neuropsychiatric symptoms; Behavioral and Psychological Symptoms of Dementia; Neuromodulation; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Alzheimer Disease; Depression; Behavior | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active stimulation (Active Comparator): Duration: 30 minutes Intensity: 2 mA Placement: left dorsolateral prefrontal cortex and right supraorbital area Size of electrodes: 5 cm x 7 cm Frequency: 5 days a week for three weeks
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham stimulation (Sham Comparator): Duration: 30 minutes Intensity: 2 mA Placement: left dorsolateral prefrontal cortex and right supraorbital area Size of electrodes: 5 cm x 7 cm Frequency: 5 days a week for three weeks
  Interventions: Other: Sham Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation
  Arms: Active stimulation
Other: Sham Stimulation
  Arms: Sham stimulation

SUMMARY:
This project will investigate the safety and efficacy of transcranial direct current stimulation (tDCS) in the treatment of depression among patients with Alzheimer's disease. The investigators aim to ameliorate depressive symptoms among patient with Alzheimer's disease, by anodal stimulation on left dorsolateral prefrontal cortex and cathodal suppression on right supraorbital area. Active stimulation will be compare to sham condition in 20 patients (10 in each groups).

DETAILED DESCRIPTION:
This project will investigate the safety and efficacy of transcranial direct current stimulation (tDCS) in the treatment of depression among patients with Alzheimer's disease. tDCS causes an excitatory effect on the anode side and suppressing effect on the cathode side through sculp with very week currents (2 mA in this project). The investigators aim to ameliorate depressive symptoms among patient with Alzheimer's disease, by anodal stimulation on left dorsolateral prefrontal cortex and cathodal suppression on right supraorbital area. Active stimulation will be compare to sham condition in 20 patients (10 in each groups) from outpatient clinic in National Center of Neurology and Psychiatry, Japan.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who meets criteria of probable Alzheimer's disease defined by NINCDS-ADRDA research criteria.
2. Participants who meets criteria of depression in Alzheimers defined by NIMH criteria.
3. Participants who have been on fixed dose (including participants without any prescription) of antidepressants for at least two weeks on the screening visit.
4. Participants who have been on fixed dose (including participants not prescribed) of antidementia drugs (donepezil, rivastigmine, galantamine, and memantine) for at least for weeks on the screening visit.
5. Ambulatory participants with or without any aiding device
6. Participants who have one caregiver, who must live with the patient at least ten hours a week and must report the patient's behavior.
7. A study partner who can report how the participant is doing is needed.
8. Eligible family member must sign and give consent on behalf of participants, whereas participants can give assent.

Exclusion Criteria: Following potential participants will be excluded

1. In case their cognitive deficits are better explained by another disease (e.g., cerebral infarction, Parkinson disease, multiple sclerosis, normotensive hydrocephalus).
2. In case they have history of epilepsy
3. In case they need treatment by antipsychotics due to significant psychotic symptoms
4. In case they have urgent risk of suicide or severe depression and any doctor require their hospitalization to psychiatric units.
5. In case they have history of ineffectiveness with electroconvulsive therapy (ECT) or transcranial direct current stimulation (tDCS)
6. In case ECT or tDCS is clinically contraindicated
7. In case they are taking benzodiazepines or antiepileptic drugs on the screening visit
8. In case they scored less than ten on Mini Mental State Exam (MMSE) or scored 3 or more on Clinical Dementia Rating (CDR)
9. In case his/her GDS score is lower than 6 at baseline
10. In case he/she is unable to agree video recording on evaluation interview

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-12; Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Attrition rate due to any adverse event | three weeks

SECONDARY OUTCOMES:
Rate of adverse events related to tDCS procedure | three weeks
Geriatric Depression Scale | one week, two weeks, three weeks, five weeks (followup)
  a subjective scale for depressive symptoms
Cornell Scale for Depression in Dementia | two weeks, three weeks, five weeks (followup)
  a objective scale for depressive symptoms
Neuropsychiatric Inventory | three weeks, five weeks (followup)
  a objective scale for neuropsychiatric symptoms
Zarit Burden Interview | three weeks, five weeks (followup)
  a subjective scale for caregivers' burden
Clinical Global Impression of Improvement | one, two, three and five weeks (followup)
  Clinician-rated impression of improvement
Starkstein Apathy Scale | two, three and five weeks (followup)
  a subjective scale for apathy

OTHER OUTCOMES:
Clinical Dementia Rating | baseline
  severity of dementia
Quality of Life - Alzheimer's Disease | baseline
  a QoL scale
ADCS-ADL | baseline
  Alzheimer's Disease Co-operative Study - Activity of Daily Living

CONTACTS AND LOCATIONS:
Overall Officials: Yuma Yokoi, MD, Principal Investigator — National Center of Neurology and Psychiatry, Japan
Locations (1):
- National Center of Neurology and Psychiatry, Kodaira, Tokyo, Japan

REFERENCES:
- [Derived] Narita Z, Yokoi Y. Transcranial direct current stimulation for depression in Alzheimer's disease: study protocol for a randomized controlled trial. Trials. 2017 Jun 19;18(1):285. doi: 10.1186/s13063-017-2019-z. PMID 28629447
- See also: UMIN CTR database — https://upload.umin.ac.jp/cgi-open-bin/ctr/ctr.cgi?function=brows&action=brows&type=summary&recptno=R000016938&language=J